CLINICAL TRIAL: NCT05113849
Title: A Phase 1, Open-label, Dose-escalation Study to Assess the Safety, Reactogenicity, and Immunogenicity of a SARS-CoV-2 Vaccine (IN-B009) in Healthy Adults Aged at 19 to 55 Years
Brief Title: Study to Evaluate the Safety and Immunogenicity of SARS-CoV-2 Vaccine (IN-B009) in Healthy Adults (COVID-19)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IN_COV_101
Record Dates: First submitted 2021-10-29; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Low-dose group) (Experimental): IN-B009 (Low-dose)
  Interventions: Biological: IN-B009 (Low-dose)
- Cohort B (High-dose group) (Experimental): IN-B009 (High-dose)
  Interventions: Biological: IN-B009 (High-dose)

INTERVENTIONS:
Biological: IN-B009 (Low-dose) — Two doses, intramuscular injection
  Arms: Cohort A (Low-dose group)
Biological: IN-B009 (High-dose) — Two doses, intramuscular injection
  Arms: Cohort B (High-dose group)

SUMMARY:
This is a first in human, phase I, open-label, dose-escalation study to assess the safety, reactogenicity, and immunogenicity of a SARS-CoV-2 Vaccine (IN-B009) in healthy adults.

DETAILED DESCRIPTION:
Total of 40 participants will be enrolled in 3 institutions : Seoul National University Hospital, Jeonbuk National University Hospital, and Chungbuk National University Hospital.

Safety, reactogenicity, and immunogenicity will be evaluated in healthy participants with administration of IN-B009 (Injected twice, 21-day-interval).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between the ages of 18 and 55 years.
* Participants considered 'healthy' to be eligible for study participation.
* Participants who are willing and able to comply with all scheduled visits and other study procedures.
* Participants with Body mass index (BMI) within the normal range.
* Participants with deltoid muscle capable of IP injection.
* Those that agreed to using medically approved contraception.
* Female participants with potential pregnancy- Those that used medically approved contraception and has negative result at the pregnancy test.
* Capable of giving personal signed informed consent

Exclusion Criteria:

* Clinically significant symptoms prior to IP injection.
* Confirmed to be COVID-19 RT-PCR positive or to have made close contact with SARS-CoV-2 infected patient.
* History of virologically-confirmed SARS, MERS, or COVID-19.
* History of congenital or acquired immunodeficiency or autoimmune diseases.
* Positive result of hepatitis B, C, RPR test, or HIV.
* History of disorder that inhibits intramuscular injection of the vaccine.
* History of hypersensitivity and severe allergic reaction to any of the components of IP.
* History of malignant tumor within 5 years prior to the first IP injection.
* Clinically significant chronic diseases that could cause safety concerns regarding COVID-19.
* Scheduled of , or history of surgery under general anaesthesia prior to first IP injection,
* Female participant that is pregnant or is currently breastfeeding.
* Smoker or history of smoking within 12 weeks prior to first IP injection.
* Previous vaccination or treatment for prevention of COVID-19.
* Vaccination prior to the first IP injection or scheduled of vaccination after second IP injection.
* Treated with immunoglobulin and/or blood/blood components prior to first IP injection.
* Chronic use of immunosuppressant prior to first IP injection.
* Participated in other clinical study prior to first IP injection, or scheduled to participate in other study during the study period.
* Healthcare worker or emergency response personnel.
* Conditions that may influence the evaluation of the study objectives.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence rate of Immediate Adverse Reaction (IAR) | Through 30 minutes post each vaccination (2 hours for sentinel participants)
Occurrence rate of solicited local and systemic AE | Through Day 7 post each vaccination
Occurrence rate of unsolicited AE | Through Day 28 post each vaccination
Occurrence rate of SAEs, MAAEs, AESIs | Through Day 365 post last vaccination
GMT of Anti-SAS-CoV-2 RBD IgG measured with ELISA | Through Day 365 post last vaccination
GMFR of Anti-SAS-CoV-2 RBD IgG from baseline measured with ELISA | Through Day 365 post last vaccination
Proportion of participants achieving a greater than or equal to 4-fold rise from baseline in IgG titer | Through Day 365 post last vaccination
GMT of Neutralizing anti-SARS-CoV-2 measured with live virus neutralization assay | Through Day 365 post last vaccination
GMFR of Neutralizing anti-SARS-CoV-2 measured with live virus neutralization assay | Through Day 365 post last vaccination
Proportion of participants achieving a greater than or equal to 4-fold rise from baseline in wild-type neutralizing antibody titer | Through Day 365 post last vaccination
Cell-mediated response | Through Day 28 post last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: In Jin Jang, Principal Investigator — Seoul National University Hospital; Min Geol Kim, Principal Investigator — Jeonju National University Hospital; Jun Ki Hwang, Principal Investigator — Chungbuk National University Hospital
Locations (3):
- South Korea (3):
  - Chungbuk National University Hospital, Chungju
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul